CLINICAL TRIAL: NCT06421649
Title: An Evaluative Commissioning Study to Investigate the Role of Adjuvant Proton Beam Radiotherapy in Patients With Localised Parotid Carcinoma
Brief Title: Investigating the Role of Adjuvant Proton Beam Therapy in Patients With Parotid Carcinoma
Acronym: PRONTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp218 (01)
Record Dates: First submitted 2024-04-25; First posted 2024-05-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-05

CONDITIONS: Parotid Cancer
Keywords: proton beam therapy; protons; evaluative commissioning
MeSH Terms: conditions — Parotid Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: Evaluative commissioning study. This is a single arm, non-randomised study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Beam Therapy (Experimental): All patients will be offered radical adjuvant proton beam therapy to a dose of 60-66 Gray (Gy) in 30-33 fractions delivered Monday to Friday over 6-6.5 weeks.
  Interventions: Radiation: Proton Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — All patients will be offered radical adjuvant proton beam therapy to a dose of 60-66 Gray (Gy) in 30-33 fractions delivered Monday to Friday over 6-6.5 weeks.

SUMMARY:
Proton Beam Therapy (PBT) is an advanced radiotherapy technique. There are two National Health Service (NHS) PBT treatment centres in the UK, one in Manchester and one in London. The NHS is committed to ensuring the best use of this limited resource by investigating which patients will benefit from PBT treatment.

Evaluative Commissioning in Protons (ECIP) is a programme of studies that explore the role of PBT for patients with different types of cancer. They are funded by NHS England. ECIP studies are not randomised studies, which means that all eligible patients will be offered proton therapy. Any patient in the United Kingdom (UK) can be referred, and for patients that need to travel far to their nearest centre, accommodation will be available.

The main benefit of PBT, compared with photon radiotherapy, is the predicted reduction in radiation dose to surrounding healthy tissues. With photon radiotherapy, some radiation passes beyond the target area, affecting healthy tissues and causing side-effects. With PBT, the radiation dose stops within the target area, causing less damage to surrounding tissues, and limiting side effects.

PRONTO is a study within the ECIP programme exploring whether PBT can reduce treatment side effects for patients with salivary gland cancers who need radiotherapy following surgery. Whilst radiotherapy is associated with good cancer control, it commonly causes problematic side-effects such as loss of taste and dry mouth. These can be permanent and can negatively affect someone's quality of life. PRONTO's main aim is to see if PBT can reduce the loss of taste following radiotherapy.

Participants in PRONTO will be closely monitored by the medical team and with questionnaires. The patient experience will be compared to what we would expect with standard photon radiotherapy.

DETAILED DESCRIPTION:
Malignant parotid tumours are uncommon. Whilst 85% of salivary gland tumours originate in the parotid gland, only 20-25% of these are malignant, representing only 3-6% of head and neck cancers. This is about 650 patients/year in the UK.

Standard treatment for local disease is with surgical resection followed by adjuvant radiotherapy for patients with high-risk features. Local control and 5-year survival rates are good, at >70% and >80% respectively, but radiotherapy is associated with considerable toxicity. More than 70% of patients receiving photon therapy experience significant dysgeusia (taste loss/alteration). This can be permanent, is associated with weight loss, diminished appetite, dry mouth, and negatively impact on Quality of Life (QoL).

The putative benefit of proton beam radiotherapy (PBT) relates to its characteristic deposition in the body, which limits the radiation dose received by surrounding healthy tissues. We hypothesise that irradiating the post-operative parotid bed with PBT rather than Intensity Modulated Radiation Therapy (IMRT), will reduce the dose delivered to the Organs at Risk (OAR), in particular the oral cavity (OC), leading to a reduction in acute and long term taste loss/alteration. The advantageous physical properties of PBT may also improve other side effects including fatigue, mucositis, nausea & vomiting and potentially hearing problems, as well as overall QoL.

Radiotherapy planning studies:

Radiation planning studies have repeatedly shown statistically significant reductions in the dose delivered to healthy tissues including: the oral cavity, brainstem, spinal cord, contralateral parotid, ipsilateral and contralateral submandibular glands and ipsilateral temporal lobe. In particular, radiotherapy doses to the oral cavity are significantly reduced, typically to below 10 Gray (Gy). No routinely contoured OAR or region of interest was consistently found to have higher doses planning with protons, although skin dose may be higher.

Clinical Trials:

Whilst there are no randomised control trials comparing protons and photons for this cohort. However, there is some clinical evidence that the use of PBT leads to clinically meaningful improvements in the side effects experienced by patients. One study compared acute toxicities between matched groups receiving either protons or photons, demonstrating statistically significant reductions in dysgeusia, fatigue, mucositis and nausea and vomiting in patients undergoing proton treatment. In other studies, PBT is associated with very low toxicity level, such as less than 30% of patients experiencing any dysgeusia. This compares favourably to photon experience, such as in the phase 3 randomised controlled trial 'A Multicentre Randomised Study of Cochlear Sparing Intensity Modulated Radiotherapy Versus Conventional Radiotherapy in Patients with Parotid Tumours' (COSTAR) where approximately 60% of patients reported dysgeusia in the Head & Neck 35 (HN35) questionnaire at 1 year. The PRONTO study is powered to identify a clinically meaningful reduction in taste dysfunction of at least 20%.

Whilst late toxicities are also likely under-reported in the retrospective international data, the published literature to date is very reassuring. The mean dose to the ipsilateral temporal lobe is reportedly reduced, and reflected in low levels of subsequent headache, fatigue and/or memory change. Similarly, whilst poorly captured, low levels of hearing dysfunction or otalgia have also been reported following PBT.

There is no rationale at all that cancer outcomes, either local control or overall survival, will be worse with PBT than photon treatment. In studies to date, local control (approximately 95%) and overall survival (89%-96%) has been excellent, and comparative to known photon experience.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Histologically confirmed primary malignant tumours of parotid gland.
3. Requiring post-operative radiotherapy to the parotid bed, with a dose equivalent of at least 60 Gray (Gy) in 2 Gy / fraction.
4. Treatment delivered with radical intent.
5. All patients must be suitable to attend regular follow-up, audiograms, toxicity monitoring, and be available for long term follow-up.
6. Willingness to comply with the protocol, including travel to the proton centre for Intensity Modulated Proton Therapy (IMPT) treatment.
7. Written informed consent.

Exclusion Criteria:

1. Previous radiotherapy to the head and neck region;
2. Parotid tumours requiring primary radiation or those with gross residual disease;
3. Metastases from squamous cell carcinoma of the head and neck to the parotid gland;
4. Benign tumours requiring post operative radiotherapy;
5. Previous or concurrent illness, which in the investigators opinion would interfere with either completion of therapy or follow-up;
6. Patients requiring or receiving neoadjuvant, concomitant or planned adjuvant chemotherapy.
7. Patients who are eligible for PBT under routine commissioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Taste dysfunction | 12 months
  Taste dysfunction as recorded on the European Organisation for the Research & Treatment of Cancer (EORTC) Head & Neck 43 (HN43) patient reported questionnaire.
  43 questions with a Likert scale of 1 - 4 Higher score may mean a worse outcome

SECONDARY OUTCOMES:
Clinician reported acute and late toxicity using Common Terminology Criteria for Adverse Events (CTCAE) grades | up to 24 months
  Using the CTCAE toxicity grade Grades 1 - 5 Higher score may mean a worse outcome
Clinician reported acute and late toxicity using Late Effects Normal Tissue - Subjective Objective Management Analytic (LENT-SOMA) scale | up to 24 months
  Using the LENT-SOMA scale A multiple item scoring system composed of four domains; subjective, objective, management and analytic.
  Grades 0-4 Higher score may mean a worse outcome
Clinician reported acute and late toxicity - measurement of hearing changes | up to 24 months
  Using pure tone audiometry to measure hearing changes Loss of hearing may mean a worse outcome
Patient reported acute and late toxicity using European Organisation for the Research & Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 module questionnaire | up to 24 months
  Using the EORTC QLQ-C30 30 questions using a Likert scale of 1-4 Higher score may mean a worse outcome
Patient reported acute and late toxicity using European Organisation for the Research & Treatment of Cancer (EORTC) Head & Neck 43 (HN43) patient reported questionnaire. | up to 24 months
  Using the EORTC HN43 patient reported questionnaire 43 questions using a Likert scale of 1-4 Higher score may mean a worse outcome
Patient reported acute and late toxicity using University of Washington Quality of Life (UW-QoL) questionnaire | up to 24 months
  Using the UW-QoL questionnaire Most questions are scored on a Likert scale, 0=worst, 100=best Lower score may mean worse outcomes
Patient reported acute and late toxicity using Glasgow hearing Aid Benefit Profile (GHABP) questionnaire | up to 24 months
  Using the GHABP questionnaire Possible values for response options (0=not applicable, 5=cannot manage at all) Higher score may mean worse outcomes
Loco-regional tumour control | up to 24 months
  This will be measured as time to recurrence (measured in months from completion of treatment) and location of recurrence (within the primary nodal regional or distant spread)
Overall survival | up to 24 months
  This will be measured in months from completion of treatment to death
Patient participation in the study each year | up to 24 months
  Number of patients referred to and participating in the study annually
Study completion rates | up to 24 months
  Review the number of patients completing radiotherapy and the number of patients completing follow up on the study as per protocol.
Oral cavity radiation dose | 12 months
  Patients will be re-planned with photon radiotherapy, the dose distribution differences between the treatment proton plans and photon plans will be recorded in particular the dose to the oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nutting, Principal Investigator — Royal Marsden NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romesser PB, Cahlon O, Scher E, Zhou Y, Berry SL, Rybkin A, Sine KM, Tang S, Sherman EJ, Wong R, Lee NY. Proton beam radiation therapy results in significantly reduced toxicity compared with intensity-modulated radiation therapy for head and neck tumors that require ipsilateral radiation. Radiother Oncol. 2016 Feb;118(2):286-92. doi: 10.1016/j.radonc.2015.12.008. Epub 2016 Feb 8. PMID 26867969